CLINICAL TRIAL: NCT00759499
Title: Obtaining and Storing Wound Debridment Samples for Immediate or Future Wound-Related Scientific Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Principal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-004
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Wound
Keywords: study of debridement tissue for research purposes.; open wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The intent of this protocol is to salvage wound material that is normally destined for destruction, so it can be used in wound-related scientific studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Debridement: The intent of this protocol is to salvage wound material that is normally destined for destruction, so it can be used in wound-related scientific studies. This clinical wound material can be studied in order to better understand the molecular, cellular, or ecological components of the wound system. These studies may be able to provide important insights into the keys of wound healing, wound persistence, or wound deterioration.

SUMMARY:
Debridement Samples being collected for future or immediate research purposes.

DETAILED DESCRIPTION:
Inclusion Criteria

1. The subject must have a full thickness wound.
2. The subject must be a candidate for sharp debridement.
3. The subject must be 18 years of age or older
4. The subject must be mentally competent as determined by the Principal Investigator.

Exclusion Criteria

1. The subject may not be currently incarcerated or pregnant.

* Nursing home and hospitalized subjects will not be excluded from this study because these subjects represent a large part of the wounded population.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have a full thickness wound.
* The subject must be a candidate for sharp debridement.
* The subject must be 18 years of age or older
* The subject must be mentally competent as determined by the Principal Investigator

Exclusion Criteria:

* The subject may not be currently incarcerated or pregnant.
* Nursing home and hospitalized subjects will not be excluded from this study because these subjects represent a large part of the wounded population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified because their wound(s) possesses something of special interest. A special interest wound can include, but will not be limited to wounds that are rapidly deteriorating, wounds diagnosed as pyoderma gangrenosum, wounds showing unusually rapid wound healing, wounds with abnormal microorganisms, non-healing wounds, young wounds, and others.
Sampling Method: Probability Sample
Enrollment: 829 (Estimated)
Dates: Start 2007-01; Primary Completion 2021-01-18 (Estimated); Study Completion 2021-01-18 (Estimated)

PRIMARY OUTCOMES:
The intent of this protocol is to salvage wound material that is normally destined for destruction, so it can be used in wound-related scientific studies. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Soutwest Regional Wound Care Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No